CLINICAL TRIAL: NCT03033355
Title: A Prospective Study of Higher Neural Control Changes Following Intra-detrusor Injection of Onabotulinumtoxin-A in Patients With Multiple Sclerosis and Lower Urinary Tract Symptoms.
Brief Title: Central Nervous System Changes Following OnabotulinumtoxinA Injection in the Bladder
Status: Completed | Type: Observational
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Rose Khavari, M.D., Principal Investigator, The Methodist Hospital Research Institute
Other Study IDs: Pro00010110
Record Dates: First submitted 2016-07-15; First posted 2017-01-26 (Estimated); Results first posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Multiple Sclerosis; Lower Urinary Tract Symptoms; Neurogenic Bladder; Detrusor, Overactive; Urge Incontinence
Keywords: Neurogenic Bladder, Detrusor Overactivity, Botox, fMRI
MeSH Terms: conditions — Multiple Sclerosis; Lower Urinary Tract Symptoms; Urinary Bladder, Neurogenic; Urinary Bladder, Overactive; Urinary Incontinence, Urge | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pre and post BTX-A injection: Female patients with confirmed diagnosis of Multiple Sclerosis referred to our Neuro-urology clinic with neurogenic lower urinary tract dysfunction receiving intra-detrusor injection of onabotulinumtoxin-A.
  Interventions: Drug: Intra-detrusor injection of Onabotulinumtoxin-A

INTERVENTIONS:
Drug: Intra-detrusor injection of Onabotulinumtoxin-A — Using cystoscopy, Onabotulinumtoxin-A is injected into the bladder.
  Other Names: OnabotulinumtoxinA, Botox®

SUMMARY:
The purpose of this research study is to evaluate higher neural changes following intra-detrusor injection of Onabotulinumtoxin-A (BTX-A) in patients with Multiple Sclerosis (MS).

We will use our prospectively collected cohort of patients. Concurrent Urodynamic and Functional Magnetic Resonance (fMRI) data will be recorded pre- and post-intravesical injection of BTX-A in patients with Multiple Sclerosis (MS) and neurogenic detrusor activity (NDO).

DETAILED DESCRIPTION:
Multiple Sclerosis is a severe debilitating disease that affects patient's quality of life. Up to 90% of patients with MS will develop lower urinary tract dysfunction within the first 18 years of the disease. Lower urinary tract symptoms (LUTS) can range from urgency to urge urinary incontinence and/or hesitancy and incomplete bladder emptying. Urgency, frequency, and neurogenic detrusor overactivity (NDO) are the most common urologic findings (34-99%) during diagnostic evaluations of patients with MS. Even though anticholinergic or beta agonist drugs have limited effectiveness and adverse side effects, they are the first line pharmacotherapy for patients with NDO if behavioral modifications and pelvic floor physical therapy are unsuccessful. Onabotulinumtoxin-A (BTX-A) intra-detrusor injection is a highly effective treatment option for patients with NDO who are refractory to more conservative management. BTX-A blocks the release of acetylcholine at the neuromuscular junction and leads to a temporary chemodenervation of the bladder (paralysis of the muscle). Motor effects of BTX-A on the bladder have been extensively studied and widely reported in the literature, and the US Food and Drug Administration has approved BTX-A for the treatment of detrusor overactivity in neurogenic and non-neurogenic patients. However, the sensory effects of BTX-A injection correlating to central nervous system regional perception/localization of urgency, frequency, and urge incontinence in humans are not well known.

Over the past decades, functional MRI (fMRI) has been used to study the activation of supraspinal lower urinary tract control centers in healthy subjects during the storage and voiding phases. Given these facts, the investigators are interested in evaluating the role of intra-detrusor injection of BTX-A in afferent response in patients with MS and NDO. High-resolution neuroimaging techniques will help investigators to further understand how MS affects the bladder-brain controls. This study will use fMRI and task-related blood oxygen level dependent (BOLD) signal to evaluate patients with MS and NDO prior to, and 6-10 weeks after intra-detrusor injection of BTX-A with simultaneous urodynamic evaluation.

Clinical correlation between women with these chronic urologic problems and new discoveries at level of central nervous system activity will give a better understanding of this disorder, leading to the development of more effective diagnostic and treatment modalities.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical diagnosis of neurogenic bladder.
* History of any neurologic illness or injury (including but not limited to spinal cord injury, Multiple Sclerosis, spina bifida, Parkinson's, major spine surgery).
* 18 years or older.
* Female patients.

Exclusion Criteria:

* Male
* History of any incontinence surgery (sling, Marshall-Marchetti-Krantz Procedure, Burch).
* History of any lower urinary tract surgery or manipulation (urethral dilation).
* Positive urine pregnancy test at enrollment .

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female subjects diagnosed with Multiple Sclerosis and lower urinary tract symptoms who are refractory to conservative management for neurogenic detrusor overactivity.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rose Khavari, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- BTX-A Injection: Female patients with confirmed diagnosis of Multiple Sclerosis referred to our Neuro-urology clinic with neurogenic lower urinary tract dysfunction, receiving intra-detrusor injection of Botulinum Toxin-A.
Period: Overall Study
Arm/Group | BTX-A Injection
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patient demographics
Groups:
- BTX-A Injection: Female patients with confirmed diagnosis of Multiple Sclerosis referred to our Neuro-urology clinic with neurogenic lower urinary tract dysfunction receiving intra-detrusor injection of Onabotulinumtoxin-A.
Arm/Group | BTX-A Injection
Number analyzed (Participants) | 12
Age, Continuous [Mean (Full Range); unit: years] | 43.9 [38 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 10
  Black | 1
  Declined | 1
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Blood Oxygen Level Dependent (BOLD) Signals in the Brain After Treatment
Description: Brain activation patterns associated with the strong desire to void (Full Urge) were examined using functional magnetic resonance imaging (fMRI), assessing BOLD signal intensity in predefined regions of interest at baseline and 6-10 weeks following OnabotulinumtoxinA (OnabotA) injection. Post-treatment changes in activity (voxel signal) were analyzed based on a statistical threshold, with increased activation defined by a T-value greater than or equal to 2.0 and decreased activation by a T-value less than or equal to 2.0.
Time Frame: Baseline (pre-OnabotA) and 6-10 weeks post-OnabotA treatment
Measure: Mean (Full Range); unit: BOLD Signal Change Derived T-Value
Arm/Group | Pre and Post BTX-A Injection
Number analyzed (Participants) | 12
BOLD Signal Change Derived T-Value
  Right Cingulate Body | 2.6 [-3.9 to 3.5]
  Left Posterior Cingulate | 2.6 [-3.9 to 3.5]
  Left Anterior Cingulate | 3.5 [-3.9 to 3.5]
  Right Prefrontal Cortex | 2.6 [-3.9 to 3.5]
  Left Insula | 2.6 [-3.9 to 3.5]
  Pons Micturition Center | 2.4 [-3.9 to 3.5]
  Left Cerebellum | -3.9 [-3.9 to 3.5]
  Left Fusiform Gyrus | -3.1 [-3.9 to 3.5]
  Left Lentiform Nucleus | -2.1 [-3.9 to 3.5]
  Right Lentiform Nucleus | -2.6 [-3.9 to 3.5]
  Left Amygdala/parahippocampal Gyrus | -2.0 [-3.9 to 3.5]
Statistical Analysis 1: Comparison: Pre and Post BTX-A Injection; Right Cingulate Body; Test type: Other; p = 0.0012, Student t-Test — Threshold for statistical significance used P-value <0.05
Statistical Analysis 2: Comparison: Pre and Post BTX-A Injection; Left Posterior Cingulate; Test type: Other; p = 0.02, student t-test — Threshold for statistical significance used P-value <0.05
Statistical Analysis 3: Comparison: Pre and Post BTX-A Injection; Left Anterior Cingulate; Test type: Other; p = 0.0015, student t-test — Threshold for statistical significance used P-value <0.05
Statistical Analysis 4: Comparison: Pre and Post BTX-A Injection; Right Prefrontal Cortex; Test type: Other; p = 0.0015, student t-test — Threshold for statistical significance used P-value <0.05
Statistical Analysis 5: Comparison: Pre and Post BTX-A Injection; Left Insula; Test type: Other; p = 0.0138, student t-test — Threshold for statistical significance used P-value <0.05
Statistical Analysis 6: Comparison: Pre and Post BTX-A Injection; Pons Micturition Center; Test type: Other; p = 0.049, student t-test — Threshold for statistical significance used P-value <0.05
Statistical Analysis 7: Comparison: Pre and Post BTX-A Injection; Left Cerebellum; Test type: Other; p = 0.001, student t-test — Threshold for statistical significance used P-value <0.05
Statistical Analysis 8: Comparison: Pre and Post BTX-A Injection; Left Lentiform Nucleus; Test type: Other; p = 0.026, student t-test — Threshold for statistical significance used P-value <0.05
Statistical Analysis 9: Comparison: Pre and Post BTX-A Injection; Right Lentiform Nucleus; Test type: Other; p = 0.026, student t-test — Threshold for statistical significance used P-value <0.05
Statistical Analysis 10: Comparison: Pre and Post BTX-A Injection; Left Amygdala/parahippocampal Gyrus; Test type: Other; p = 0.015, student t-test — Threshold for statistical significance used P-value <0.05

2. Secondary Outcome: Changes in Urodynamic (UDS) Parameters Following OnabotA Treatment
Description: Objective clinical assessments examined changes in urodynamic (UDS) parameters collected during functional MRI (fMRI) sessions at baseline (pre-OnabotA) and 6-10 weeks post-treatment. These included final post-void residual (PVR) volume and maximum cystometric capacity (MCC). MCC was measured during the first bladder infusion cycle of each neuroimaging session and represents the bladder volume at which an individual can no longer delay voiding during bladder filling. An increase in MCC following OnabotA treatment may indicate improved bladder storage capacity, particularly in individuals with reduced bladder compliance or capacity. PVR reflects the volume of urine remaining in the bladder after voiding (measured in CC or mL); higher PVR values suggest less effective bladder emptying.
Time Frame: Baseline (Pre-OnabotA) and 6-10 Weeks Post-OnabotA Treatment
Measure: Mean (Full Range); unit: Cubic Centimeters
Groups:
- Pre-OnabotA UDS Parameters: The following metrics reflect the urodynamic assessments of participants before OnabotA treatment.
- Post-OnabotA UDS Parameters: The following metrics reflect the urodynamic assessments of participants following OnabotA treatment.
Arm/Group | Pre-OnabotA UDS Parameters | Post-OnabotA UDS Parameters
Number analyzed (Participants) | 12 | 12
Cubic Centimeters
  Final Post Void Residual (PVR) Volume | 261.4 [70 to 650] | 377.9 [120 to 600]
  Maximum Cystometric Capacity (MCC) During 1st fMRI/UDS Bladder Filling | 134.5 [14 to 251] | 195.5 [51 to 401]

3. Secondary Outcome: Number of Participants Presenting With Neurogenic Detrusor Overactivity (NDO) Events During Urodynamic Studies (UDS) Before and After OnabotA Treatment
Description: This outcome measure assesses the incidence of neurogenic detrusor overactivity (NDO) events observed during fMRI/UDS sessions conducted at baseline (pre-OnabotA) and 6-10 weeks following OnabotA treatment. Detrusor overactivity refers to involuntary detrusor muscle contractions observed during the bladder filling phase, which may be spontaneous or provoked. In individuals with neurogenic lower urinary tract dysfunction, these involuntary contractions are attributed to underlying neurologic conditions and are classified as NDO. The presence or absence of NDO events was determined based on detrusor pressure tracings recorded during the bladder filling phase. Participants were categorized as positive for NDO if one or more involuntary contractions were observed. A decrease in the number of participants with NDO events following OnabotA treatment suggests a therapeutic effect on detrusor overactivity and may indicate improved bladder control and reduced urgency or incontinence symptoms.
Time Frame: Baseline (Pre-OnabotA) and 6-10 Weeks Post-OnabotA Treatment
Measure: Count of Participants; unit: Participants
Groups:
- Incidence of NDO Events During UDS Pre-OnabotA: The following metrics reflect the urodynamic assessments of participants before OnabotA treatment.
- Incidence of NDO Events During UDS Post-OnabotA: The following metrics reflect the urodynamic assessments of participants following OnabotA treatment.
Arm/Group | Incidence of NDO Events During UDS Pre-OnabotA | Incidence of NDO Events During UDS Post-OnabotA
Number analyzed (Participants) | 12 | 12
Participants | 6 | 1

4. Secondary Outcome: Changes in Subjective Clinical Outcomes Following Treatment - Urogenital Distress Inventory, Short Form (UDI-6)
Description: The Urinary Distress Inventory, Short Form (UDI-6), is a validated questionnaire used to assess the severity of urinary symptoms and their impact on quality of life. It consists of six items evaluating urinary frequency, urgency-related leakage, stress-related leakage, difficulty emptying the bladder, and discomfort or pain in the lower abdomen or genital area. Each item is scored on a Likert scale (0-4), with higher scores indicating greater symptom-related distress.Total UDI-6 scores are calculated by adding all 6 questions with scores ranging from 0 to 24, where higher scores indicate worse symptoms.
  In this study, we report overall UDI-6 total scores (range: 0-24) as well as individual scores (range:0-4) for Questions 1 (urinary frequency) and 2 (urge urinary incontinence) at two timepoints: baseline (pre-OnabotA) and 6-10 weeks following OnabotA treatment.
Time Frame: Baseline (Pre-OnabotA) and 6-10 Weeks Post-OnabotA Treatment
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Pre-OnabotA Validated Questionnaire Scores: The following metrics reflect patient reported validated symptom scores before OnabotA treatment.
- Post-OnabotA Validated Questionnaire Scores: The following metrics reflect patient reported validated symptom scores following OnabotA treatment.
Arm/Group | Pre-OnabotA Validated Questionnaire Scores | Post-OnabotA Validated Questionnaire Scores
Number analyzed (Participants) | 12 | 12
score on a scale
  Total UDI-6 Score | 12.09 [6 to 21] | 6.27 [0 to 15]
  UDI-6, Q1 (Frequency) | 3.27 [2 to 4] | 1.55 [0 to 4]
  UDI-6, Q2 (Urge Urinary Incontinence) | 2.64 [0 to 4] | 1.1 [0 to 4]

5. Secondary Outcome: Changes in Subjective Clinical Outcomes Following Treatment - Incontinence Impact Questionnaire Short Form (IIQ-7)
Description: The Incontinence Impact Questionnaire Short Form (IIQ-7) is a seven-item questionnaire used to assess the impact of urinary incontinence on a person's quality of life. Each question has the following score range: 0-3 (with the highest score associated with higher symptom distress). Here we report the average overall score, which is calculated by adding scores from all 7 questions. Total score ranges from 0 to 21, with higher scores reflecting worse symptoms.
Time Frame: Baseline (Pre-OnabotA) and 6-10 Weeks Post-OnabotA Treatment
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Pre-OnabotA Validated Questionnaire Scores | Post-OnabotA Validated Questionnaire Scores
Number analyzed (Participants) | 12 | 12
score on a scale | 9.64 [0 to 18] | 4.36 [0 to 15]

6. Secondary Outcome: Changes in Voiding Diary Metrics - Urge Urinary Incontinence (UUI) Events Per Day
Description: Voiding diary entries recorded that measure the number of urge urinary incontinence (UUI) events per day. Recorded timepoints (Pre- and Post-OnabotA treatment). Measures are reported by participants that fill out voiding diaries at baseline (pre-) and post-OnabotA treatment timepoints.
Time Frame: Baseline (Pre-OnabotA) and 6-10 Weeks Post-OnabotA Treatment
Measure: Mean (Full Range); unit: Average events per day
Groups:
- Pre-OnabotA Voiding Diary Metric: The following metrics reflect the urodynamic assessments of participants before OnabotA treatment.
- Post-OnabotA Voiding Diary Metric: The following metrics reflect the urodynamic assessments of participants following OnabotA treatment.
Arm/Group | Pre-OnabotA Voiding Diary Metric | Post-OnabotA Voiding Diary Metric
Number analyzed (Participants) | 12 | 12
Average events per day | 1.64 [0 to 4] | 0.42 [0 to 1]

7. Secondary Outcome: Changes in Voiding Diary Metrics - Number of Participants Requiring Clean Intermittent Catheterization(CIC)
Description: Analysis of voiding diary metric measuring the number of participants that utilized clean intermittent catheterization (CIC) to empty their bladder. These measures were recorded at both baseline (pre-) and post-OnabotA treatment timepoints.
Time Frame: Baseline (Pre-OnabotA) and 6-10 Weeks Post-OnabotA Treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-OnabotA UDS Parameters | Post-OnabotA UDS Parameters
Number analyzed (Participants) | 12 | 12
Participants | 8 | 11

ADVERSE EVENTS:
Time Frame: Throughout the entire study (2 months)
Arm/Group | Pre and Post BTX-A Injection
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-20): https://cdn.clinicaltrials.gov/large-docs/55/NCT03033355/Prot_SAP_000.pdf